CLINICAL TRIAL: NCT04405154
Title: A Phase II Study of Concomitant Camrelizumab With Chemoradiation for Locally Advanced, Unresectable Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Concomitant Camrelizumab With Chemoradiation for Locally Advanced Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yan Li, MD, PhD, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP18-TCR-XN001
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck; Squamous Cell Carcinoma; Immune Checkpoint Inhibitors; Chemoradiation
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — camrelizumab; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Arm (Experimental): Camrelizumab every 2 weeks in combination with 6-7 weeks of radiation therapy and every 3 weeks cisplatin.
  Interventions: Biological: Camrelizumab; Drug: Cisplatin; Radiation: IMRT or VMAT

INTERVENTIONS:
Biological: Camrelizumab — Administered as an intravenous (IV) infusion every 2 weeks (Q2W): 14 days prior to radiation, then Day 1 of radiation and then every 14 days for total 8 doses.
  Other Names: SHR-1210
Drug: Cisplatin — 75-100 mg/m^2 administered as an IV infusion Q3W, for a total of 3 doses, at the same time as radiation: Day 1, Day 22, Day 43 of radiation.
  Other Names: Platinol
Radiation: IMRT or VMAT — 66-70 Gy given in 33-35 fractions over 6-7 weeks.

SUMMARY:
The goal of this study is to determine the efficacy and safety of camrelizumab given concomitantly with chemoradiation in participants with unresectable, locally advanced head and neck squamous cell carcinoma (LA-HNSCC). All participants will receive camrelizumab in addition to chemoradiation, the standard treatment for LA-HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Has a pathologically proven new diagnosis of head and neck squamous cell carcinoma
* Has unresectable disease and is eligible for definitive chemoradiation based on investigator decision
* Has Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Has evaluable tumor burden (measurable and/or non-measurable tumor lesions) based on RECIST version 1.1
* Has adequate organ function as defined
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study therapy
* Female and male participants of reproductive potential must agree to use adequate contraception throughout the study period and for up to 180 days after the last dose of study therapy

Exclusion Criteria:

* Has cancer outside of the oropharynx, larynx, and hypopharynx or oral cavity, such as nasopharyngeal, sinus, other para-nasal, or other unknown primary head and neck cancer
* Is currently participating or has participated in a study with an investigational agent or using an investigational device within 4 weeks of the first dose of study therapy
* Has history of a diagnosed and/or treated hematologic or primary solid tumor malignancy, unless in remission for at least 5 years prior to randomization
* Has a history of severe hypersensitivity reaction to camrelizumab, Cisplatin or radiotherapy
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody or has previously participated in clinical studies with camrelizumab
* Has received a live vaccine within 30 days prior to the first dose of study therapy
* Has had prior systemic therapy, targeted therapy, radiotherapy treatment or radical surgery for head and neck cancer under study
* Has not recovered from major surgery prior to starting study therapy
* Has known active Hepatitis B or C
* Has known history of Human Immunodeficiency Virus (HIV)
* Has a significant cardiovascular disease
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment
* Has had previous allogeneic tissue/solid organ transplant
* Has active infection requiring systemic therapy
* Is pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  The number of participants with radiologically confrmed complete or partial response according to RECIST 1.1

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  OS is the time from randomization to death due to any cause.
Disease-free Survival (DFS) | Up to 5 years
  DFS is the time from the date of randomization to the date of first record of disease recurrence or death.
Acute Adverse Events (AEs) | Up to 6 months
  The number of participants who experience unacceptable toxicity during protocol treatment as measured by the NCI CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, MD,PhD, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No